CLINICAL TRIAL: NCT02723669
Title: Open Label, Randomized, Two-Arm, Single-Dose, Two-Period, Crossover Study to Determine the Relative Bioavailability of AR10 (Acetylcysteine Effervescent Tablets) Compared to Reference Product in Healthy, Adult Subjects, Fasting
Brief Title: Relative Bioavailability of AR10 Compared to Reference Product
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AR10.001
Record Dates: First submitted 2016-03-17; First posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Relative Bioavailability
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AR10 (Experimental): AR10 acetylcysteine effervescent tablets for oral solution (two 0.5 g and four 2.5 g)
  Interventions: Drug: AR10
- acetylcysteine (Active Comparator): acetylcysteine solution; oral 20% (200 mg/mL)
  Interventions: Drug: acetylcysteine

INTERVENTIONS:
Drug: AR10 — effervescent tablet
  Other Names: acetylcysteine
  Arms: AR10
Drug: acetylcysteine — oral solution
  Other Names: reference product
  Arms: acetylcysteine

SUMMARY:
This study evaluates the relative bioavailability of Acetylcysteine Effervescent Tablets (AR10) and Reference N-acetylcysteine. Patients will receive both products in an Open Label, Randomized, Two-Arm, Single-Dose, Two-Period, Crossover design.

DETAILED DESCRIPTION:
An Open Label, Randomized, Two-Arm, Single-Dose, Two-Period, Crossover Study Relative Bioavailability Study. The present study is intended to compare and evaluate the relative bioavailability of a single 11 gram dose of AR10 (acetylcysteine effervescent tablets for oral solution (two 0.5 g and four 2.5 g]), and the reference Listed Drug (acetylcysteine solution; oral 20% [200 mg/mL] of American Pharmaceutical Partners) in healthy adult, human subjects under fasting conditions. A balanced block randomization schedule will be generated before the start of dosing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (males or females) between 18 - 50 years of age inclusive.
* Body weight at least 154 pounds (70 kg) and a Body Mass Index no greater than 30 kg/m2.
* Healthy as determined by medical history, clinical examination, and laboratory examination performed within 30 days prior to admission for the first period of the study.
* Subjects willing and able to provide a written informed consent, HIPPA and to adhere to the protocol requirements.
* If female and of childbearing potential (defined as a pre-menopausal female who is biologically capable of becoming pregnant), the subject must agree to remain abstinent or practice a medically acceptable form of contraception from screening until the close out visit of the clinical study. Acceptable forms of contraception include intrauterine devices, implantable devices, and barrier methods. If a barrier method is chosen, a double barrier (e.g., condom plus foam) is required.
* Negative beta human chorionic gonadotropin test, consistent with no pregnancy (females only).
* Non-smokers

Exclusion Criteria:

* Known hypersensitivity, allergy, idiosyncratic reaction or adverse reaction to acetylcysteine, its excipients, and other related compounds with similar chemical characteristics or any severe allergic reaction to any drug or multiple food/drug allergies.
* History or current evidence of clinically significant medical condition including, but not limited to, hepatic, renal, cardiac, vascular, gastrointestinal, or thyroid disease, diabetes, epilepsy, respiratory or hematological disease, acute narrow angle glaucoma, or psychiatric disorder that, in the opinion of the Principal Investigator, would confound the study results or present a risk to the subject.
* Subjects are to be without symptoms of nausea and/or vomiting. Subjects with a history of chronic nausea/vomiting are excluded. Subjects who had an acute illness/condition and have not had any nausea and/or vomiting episodes in the past two weeks may be screened provided they are medically cleared from the acute illness/condition involving nausea and/or vomiting episode(s).
* Existence of any surgical or medical condition that in the judgment of Principal Investigator might interfere with the absorption, distribution, metabolism, or elimination of the investigational product.
* Any clinically significant abnormality in the electrocardiogram (12 lead ECG).
* Laboratory values that are considered clinically significant (clinical chemistry, hematology, coagulation, urinalysis, or pregnancy test) - Note: In the event of any parameter lying outside of the normal range, the sample may be repeated once. This value will be accepted if it lies within the normal range.
* Consumption of grapefruit juice/grapefruit within 14 days prior to Period I admission.
* Use of alcohol or caffeine containing products within 72 hours of each dose of °History or presence of alcoholism or drug abuse within 1 year of study participation.
* Known or suspected carcinoma.
* Presence of the disease markers of the human immunodeficiency virus (HIV) 1 or 2, and hepatitis B or C viruses.
* Positive serum test for drug(s) of abuse testing (amphetamines, barbiturates, benzodiazepines, tetrahydrocannabinol, morphine, and cocaine, and alcohol).
* History of intake/administration of any investigational treatment in a clinical study within the last 30 days prior to the onset of the study admission in Period I.
* History of significant blood loss (≥ 350 mL) due to any reason, including blood donation, within the last 12 weeks prior to admission in Period I of the study.
* Intake/administration of any enzyme-modifying drugs or drugs that might increase or decrease acetylcysteine levels within 30 days of investigational product administration, or over-the-counter (OTC) drugs including vitamins and natural supplements within 21 days of the first dose of Investigational Product administration and throughout study unless approved by the Principal Investigator or Sponsor.
* Requirement of special diet preventing consumption of standard, healthy meals during the in-clinic portions of the study. In such cases, subject selection will be at the discretion of the Principal Investigator in discussion with Medical Monitor, if required.
* Any subject who, in the opinion of the Principal Investigator, cannot or may not follow instructions.
* Difficulty in swallowing a liquid solution.
* Female subjects with a self-reported history of anemia during menstrual cycle which may coincide with any of the dosing day(s) during the study period.
* Pregnant and lactating females.
* Employee of the Sponsor, Clinical site, or Clinical research organization.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Comparison of Area Under the Curve (AUC) profiles of the two formulations of acetylcysteine to determine the Relative Bioavailability | 10 days
  To compare AUC of a single 11 gram dose of AR10 acetylcysteine effervescent tablets for oral solution (two 0.5 g and four 2.5 g), and the Reference Listed Drug (acetylcysteine solution; oral 20% [200 mg/mL] from American Pharmaceutical Partners) in a minimum of 24 healthy adult, human subjects under fasting conditions, to establish relative bioavailability.
Comparison of Maximum Plasma Concentration (Cmax) profiles of the two formulations of acetylcysteine to determine the Relative Bioavailability | 10 days
  To compare Cmax of a single 11 gram dose of AR10 acetylcysteine effervescent tablets for oral solution (two 0.5 g and four 2.5 g), and the Reference Listed Drug (acetylcysteine solution; oral 20% [200 mg/mL] from American Pharmaceutical Partners) in a minimum of 24 healthy adult, human subjects under fasting conditions, to establish relative bioavailability.

SECONDARY OUTCOMES:
The safety and tolerability of AR10 and the reference product, as measured by treatment-emergent adverse events (AEs), concomitant medications, vital signs (pulse, temperature and respiratory rate), and assessment of well-being. | 12 days
  To compare the safety and tolerability of AR10 and the reference product, as measured by treatment-emergent adverse events (AEs), concomitant medications, vital signs (pulse, temperature and respiratory rate), and assessment of well-being.

OTHER OUTCOMES:
Evaluation of subject preference between AR10 and the reference product using the adapted British Nutritional Foundation's Sensory Evaluation (2004) 5-point hedonic scale. | 10 days
  Following each dose, subjects were asked to rate the taste, smell, flavor, texture, and overall preference of each product using the adapted British Nutritional Foundation's Sensory Evaluation (2004) 5-point hedonic scale, ranging from dislike very much to like very much. After the second dose was taken, subjects were also asked to choose which treatment they would prefer.
Evaluation of healthcare provider preference between AR10 and the reference product using the adapted British Nutritional Foundation's Sensory Evaluation (2004) 5-point hedonic scale | 10 days
  Healthcare providers involved in dispensing, preparing, and administering the study drug responded to the preference survey within 30 minutes of completing dosing activities in each study period.

CONTACTS AND LOCATIONS:
Overall Officials: Tania D Johnson, RN, BSN, Study Director — Arbor Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greene SC, Noonan PK, Sanabria C, Peacock WF. Effervescent N-Acetylcysteine Tablets versus Oral Solution N-Acetylcysteine in Fasting Healthy Adults: An Open-Label, Randomized, Single-Dose, Crossover, Relative Bioavailability Study. Curr Ther Res Clin Exp. 2016 Jun 27;83:1-7. doi: 10.1016/j.curtheres.2016.06.001. eCollection 2016. PMID 27668024